CLINICAL TRIAL: NCT02649192
Title: A Double-Blind, Randomized, Placebo-Controlled Study of Antibody Induction by Vitamin Supplementation at the Time of Influenza Virus Vaccinations in Children
Brief Title: Influenza Virus Vaccine Plus Vitamin A and D Supplements for Prevention of Respiratory Virus Infections in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLUVIT
Record Dates: First submitted 2016-01-06; First posted 2016-01-07 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Healthy Participants
Keywords: Children; Vitamin Supplements; Influenza virus vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Fumigant 93; Dietary Supplements; Medication Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Influenza Virus Vaccine Plus Vitamins A and D (Active Comparator): Participants receive influenza virus vaccine and Vitamins A and D supplement on Day 0 and Day 28.
  Interventions: Biological: Influenza virus vaccine; Dietary Supplement: Vitamins A and D
- Influenza Virus Vaccine Plus Placebo (Placebo Comparator): Participants receive influenza virus vaccine and matched placebo on Day 0 and Day 28.
  Interventions: Biological: Influenza virus vaccine; Other: Placebo

INTERVENTIONS:
Biological: Influenza virus vaccine — Children will have the first influenza virus vaccine dose (dose 1) administered on day 0 of the trial, and the second dose (dose 2) administered 28 days later.
  Other Names: Fluzone®
Dietary Supplement: Vitamins A and D — The chewable gummy contains either Vitamin A (20,000 International Units) and Vitamin D3 (2,000 International Units), which should be fully chewed under supervision of study staff with documentation in the participant's research record and eMAR (electronic medical administration record). The chewable gummy should be administered prior to receiving influenza virus vaccination.
  Other Names: Nutritional Supplement
  Arms: Influenza Virus Vaccine Plus Vitamins A and D
Other: Placebo — The chewable gummy matched placebo will be formulated with gelatin base and tangerine oil and match the Vitamin A and D in shape, taste, texture, and appearance. Gummies should be fully chewed under supervision of study staff with documentation in the participant's research record and eMAR (electronic medical administration record). The chewable gummy should be administered prior to receiving influenza virus vaccination.
  Other Names: Look-alike Medication; Matched Placebo
  Arms: Influenza Virus Vaccine Plus Placebo

SUMMARY:
Children are particularly vulnerable to respiratory virus infections, especially influenza. Vitamin A & D deficiencies are associated with vulnerability to infectious diseases of the respiratory tract. The central hypothesis of this protocol is that vitamin supplements will enhance antibody responses toward the flu vaccine in children. Children, 2-8 years old, will be randomized to receive influenza virus vaccine with a vitamin A+D supplement or influenza virus vaccine with placebo. Children will be tested for vitamin levels and immune responses before and after influenza virus vaccinations to determine if vitamin supplementation improves the influenza virus vaccine-induced immune response.

PRIMARY OBJECTIVE:

* To assess the vaccine-induced and total antibody (including IgG and IgA) response after influenza virus vaccine administration and IgA/IgG plus IgA/IgM ratios at 28 and 56 days in sera

SECONDARY OBJECTIVE:

* To assess the neutralizing response toward influenza virus vaccine in the sera.

DETAILED DESCRIPTION:
Participants will be randomized to receive either an influenza virus vaccine plus Vitamins A & D or an influenza virus vaccine plus placebo. They will be stratified based on retinol binding protein (RBP) levels at screening, using a cut-off indicative of Vitamin A insufficiency (≤22,000 ng/ml). Co-enrolled sibling participants will be first stratified by RBP levels, then siblings within the same stratum will be equally assigned to different arms to provide greater assurance of balanced treatment assignment. Children will be tested for vitamin levels and immune responses before and after influenza virus vaccinations to determine if vitamin supplementation improves the influenza virus vaccine-induced antibody immune response.

All participants will receive two doses of an influenza virus vaccination administered at least 28 days apart. Vitamin levels and antibody responses toward the vaccine will be measured on day 0 (baseline levels obtained where day 0 equals the first influenza virus vaccination administration), day 28, and day 56. Placebo or Vitamins A + D (at the levels of 20,000 IU and 2,000 IU, respectively) will be administered orally on the days of vaccination.

Blood serum samples will be collected from participants on Day 0, prior to receiving influenza virus vaccine on Day 28, and during their Day 56 follow-up visit.

Parents will be asked to fill out diary cards to indicate food intake for children during the study period along with an optional food frequency questionnaire given on day 56. Specific measurements on days 28, and 56 will include analyses of vaccine-specific and total IgA, IgG, and IgA/IgG plus IgA/IgM ratios in sera. Functional activities of antibodies toward influenza vaccine will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Resident of the Memphis area community.
* Parent or legal guardian willing and able to give informed consent and comply with study requirements.

Exclusion Criteria:

* Current use of investigational or immunosuppressive drugs (e.g., steroids) at the time of enrollment.
* Currently taking a daily (routine) vitamin A, D, or multivitamin. Note: participants who report occasional or sporadic vitamin use will be allowed to enroll.
* History of lung disease, asthma, immunodeficiency, sickle cell disease, or any other serious underlying condition or disease in the opinion of the principal investigator.
* Evidence of developmental delay or evolving neurological disorders at screening. Current use of antibiotics or antivirals at enrollment.
* History of having a severe allergy to eggs or to any inactive ingredient in the influenza virus vaccine
* History of a life-threatening reaction to influenza vaccinations
* Currently wheezing at the time of enrollment
* History of heart, kidney, or lung conditions
* History of diabetes
* Use of an anti-influenza medication (including amantadine, rimantadine, oseltamivir, and zanamivir) within 14 days prior to enrollment
* Acute febrile [>100.0°F (37.8°C) oral] illness or acute respiratory illness (e.g., cough or sore throat) within 3 days prior to enrollment
* Previous receipt of current seasonal influenza vaccine

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nehali Patel, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Groups:
- A&D - S1: Participants receiving influenza virus vaccine plus vitamin A and D supplements in 2015-16 season
- Placebo - S1: Participants receiving influenza virus vaccine plus matched placebo in 2015-16 season
- A&D - S2: Participants receiving influenza virus vaccine plus vitamin A and D supplements in 2016-17 season
- Placebo - S2: Participants receiving influenza virus vaccine plus matched placebo in 2016-17 season
- A&D - S3: Participants receiving influenza virus vaccine plus vitamin A and D supplements in 2017-18 season
- Placebo - S3: Participants receiving influenza virus vaccine plus matched placebo in 2017-18 season
Period: Overall Study
Arm/Group | A&D - S1 | Placebo - S1 | A&D - S2 | Placebo - S2 | A&D - S3 | Placebo - S3
Started | 5 | 4 | 22 | 22 | 12 | 14
Vitamin A Sufficiency (RBP≥22,000 ng/ml) | 2 | 2 | 11 | 12 | 7 | 8
Vitamin A Insufficiency (RBP<22,000 ng/m | 3 | 2 | 11 | 10 | 5 | 6
Completed | 5 | 4 | 21 | 20 | 11 | 14
Not Completed | 0 | 0 | 1 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- A&D-S1: Participants receiving influenza virus vaccine plus vitamin A and D supplements in 2015-16 season
- Total: Total of all reporting groups
Arm/Group | A&D-S1 | Placebo - S1 | A&D - S2 | Placebo - S2 | A&D - S3 | Placebo - S3 | Total
Number analyzed (Participants) | 5 | 4 | 22 | 22 | 12 | 14 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 4 | 22 | 22 | 12 | 14 | 79
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 7 [4 to 8] | 3.5 [2 to 5] | 5 [4 to 8] | 4 [2 to 8] | 3 [2 to 8] | 5 [2 to 8] | 5 [2 to 8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 14 | 14 | 6 | 6 | 46
  Male | 2 | 1 | 8 | 8 | 6 | 8 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ethnicity: Not Hispanic or Latino | 5 | 4 | 21 | 22 | 12 | 14 | 78
  Ethnicity: Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black | 5 | 4 | 15 | 16 | 8 | 9 | 57
  Race: White | 0 | 0 | 7 | 6 | 4 | 5 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 22 | 22 | 12 | 14 | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Positive Responses in Virus-specific Antibody in Sera
Description: The percentage of 2X increases or conversion from undetectable to detectable response in virus-specific antibody toward any vaccine component after 2 immunizations in intervention and control groups will be reported.
Time Frame: Day 56 after vaccination
Population: All enrolled subjects who satisfied the inclusion/exclusion criteria were included in the analysis. For the four participants who didn't complete the study, results after one immunization were used.
Measure: Number; unit: percentage of participants
Arm/Group | A&D - S1 | Placebo - S1 | A&D - S2 | Placebo - S2 | A&D - S3 | Placebo - S3
Number analyzed (Participants) | 5 | 4 | 22 | 22 | 12 | 14
percentage of participants | 80 | 75 | 100 | 100 | 100 | 100

2. Primary Outcome: Isotype Ratios on Day 56
Description: Isotype ratios will be summarized with descriptive statistics.
Time Frame: Day 56 after vaccination
Population: Subjects with complete isotype data at day 56. Subjects with an undetermined assay result were not included in analyses. In some cases, the limit of detection (LOD) for the assay was reached and that LOD value was used in calculations.
Measure: Median (Full Range); unit: ratio
Arm/Group | A&D-S1 | Placebo - S1 | A&D - S2 | Placebo - S2 | A&D - S3 | Placebo - S3
Number analyzed (Participants) | 5 | 4 | 20 | 20 | 11 | 14
ratio
  IgA/IgG1 | 0.4 [0.06 to 0.67] | 0.3 [0.22 to 0.5] | 0.3 [0.004 to 0.63] | 0.27 [0.13 to 0.47] | 0.21 [0.13 to 0.65] | 0.28 [0.12 to 0.87]
  IgA/IgG2 | 0.71 [0.24 to 0.85] | 0.69 [0.49 to 1.93] | 0.96 [0.004 to 6.3] | 1.13 [0.58 to 4.45] | 0.65 [0.19 to 2.03] | 0.75 [0.22 to 2.39]
  IgA/IgG3 | 2.73 [0.38 to 7.75] | 3.03 [1.55 to 7.44] | 1.44 [0.02 to 6.97] | 1.68 [0.29 to 5.13] | 2.4 [0.89 to 12.5] | 3.02 [0.41 to 12.3]
  IgA/IgM | 2.48 [0.16 to 2.8] | 1.37 [0.83 to 2.89] | 1.21 [0.03 to 3.06] | 1.21 [0.45 to 2.88] | 0.86 [0.23 to 1.9] | 1 [0.14 to 3.26]
Statistical Analysis 1: Comparison: A&D-S1 vs Placebo - S1; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG1 at day 56 in 2015-16 season; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: A&D - S2 vs Placebo - S2; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG1 at day 56 in 2016-17 season; Test type: Superiority; p = 0.49, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: A&D - S3 vs Placebo - S3; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG1 at day 56 in 2017-18 season; Test type: Superiority; p = 0.50, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: A&D-S1 vs Placebo - S1; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG2 at day 56 in 2015-16 season; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: A&D - S2 vs Placebo - S2; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG2 at day 56 in 2016-17 season; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: A&D - S3 vs Placebo - S3; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG2 at day 56 in 2017-18 season; Test type: Superiority; p = 0.65, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: A&D-S1 vs Placebo - S1; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG3 at day 56 in 2015-16 season; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: A&D - S2 vs Placebo - S2; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG3 at day 56 in 2016-17 season; Test type: Superiority; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: A&D - S3 vs Placebo - S3; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgG3 at day 56 in 2017-18 season; Test type: Superiority; p = 0.54, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: A&D-S1 vs Placebo - S1; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgM at day 56 in 2015-16 season; Test type: Superiority; p = 0.90, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: A&D - S2 vs Placebo - S2; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgM at day 56 in 2016-17 season; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: A&D - S3 vs Placebo - S3; Null hypothesis: No difference between intervention and placebo groups in the ratio of IgA/IgM at day 56 in 2017-18 season; Test type: Superiority; p = 0.34, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Percentage of Participants With Seroconversion at Day 56 After Vaccination, Overall
Description: Secondary analyses will examine sero-conversion based on antibody functions (HAI or neutralization) defined as antibody titers of <1:40 converting to ≥1:40, or a four-fold increase in titer for participants with a starting titer of ≥1:40. Sero-conversion rate (expressed as percentage) will be estimated with 95% confidence interval. The rate difference will be described with point estimate and 95% confidence interval.
Time Frame: Day 56 after vaccination
Population: Subjects with complete HAI data at day 56. Subjects without a day 56 sample were not included in analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | A&D-S1 | Placebo - S1 | A&D - S2 | Placebo - S2 | A&D - S3 | Placebo - S3
Number analyzed (Participants) | 5 | 4 | 21 | 20 | 11 | 14
percentage of participants
  H1N1 | 0 [0 to 0] | 0 [0 to 0] | 71.4 [47.8 to 88.7] | 95.0 [75.1 to 99.9] | 72.7 [39.0 to 94.0] | 85.7 [57.2 to 98.2]
  H3N2 | 40.0 [5.3 to 85.3] | 50.0 [6.8 to 93.2] | 71.4 [47.8 to 88.7] | 80.0 [56.3 to 94.3] | 72.7 [39.0 to 94.0] | 50.0 [23.0 to 77.0]
  B/Phuket | 0 [0 to 0] | 0 [0 to 0] | 28.6 [11.3 to 52.2] | 55.0 [31.5 to 76.9] | 45.5 [16.7 to 76.6] | 28.6 [8.4 to 58.1]
  B/Brisbane | 0 [0 to 0] | 0 [0 to 0] | 28.6 [11.3 to 52.2] | 55.0 [31.5 to 76.9] | 27.3 [6.0 to 61.0] | 35.7 [12.8 to 64.9]
Statistical Analysis 1: Comparison: A&D-S1 vs Placebo - S1; H1N1; Test type: Superiority; Treatment Difference in Seroconversion R = 0, 95% CI 2-sided [0 to 0] — Treatment group minus placebo
Statistical Analysis 2: Comparison: A&D - S2 vs Placebo - S2; H1N1; Test type: Superiority; Treatment Difference in Seroconversion R = -23.6, 95% CI 2-sided [-51.7 to 6.2] — Treatment group minus placebo
Statistical Analysis 3: Comparison: A&D - S3 vs Placebo - S3; H1N1; Test type: Superiority; Treatment Difference in Seroconversion R = -13.0, 95% CI 2-sided [-49.4 to 26.5] — Treatment group minus placebo
Statistical Analysis 4: Comparison: A&D-S1 vs Placebo - S1; H3N2; Test type: Superiority; Treatment Difference in Seroconversion R = -10.0, 95% CI 2-sided [-70.1 to 56.1] — Treatment group minus placebo
Statistical Analysis 5: Comparison: A&D - S2 vs Placebo - S2; H3N2; Test type: Superiority; Treatment Difference in Seroconversion R = -8.6, 95% CI 2-sided [-38.8 to 20.6] — Treatment group minus placebo
Statistical Analysis 6: Comparison: A&D - S3 vs Placebo - S3; H3N2; Test type: Superiority; Treatment Difference in Seroconversion R = 22.7, 95% CI 2-sided [-17.5 to 57.9] — Treatment group minus placebo
Statistical Analysis 7: Comparison: A&D-S1 vs Placebo - S1; B/Phuket; Test type: Superiority; Treatment Difference in Seroconversion R = 0, 95% CI 2-sided [0 to 0] — Treatment group minus placebo
Statistical Analysis 8: Comparison: A&D - S2 vs Placebo - S2; B/Phuket; Test type: Superiority; Treatment Difference in Seroconversion R = -26.4, 95% CI 2-sided [-54.1 to 5.8] — Treatment group minus placebo
Statistical Analysis 9: Comparison: A&D - S3 vs Placebo - S3; B/Phuket; Test type: Superiority; Treatment Difference in Seroconversion R = 16.9, 95% CI 2-sided [-23.1 to 53.3] — Treatment group minus placebo
Statistical Analysis 10: Comparison: A&D-S1 vs Placebo - S1; B/Brisbane; Test type: Superiority; Treatment Difference in Seroconversion R = 0, 95% CI 2-sided [0 to 0] — Treatment group minus placebo
Statistical Analysis 11: Comparison: A&D - S2 vs Placebo - S2; B/Brisbane; Test type: Superiority; Treatment Difference in Seroconversion R = -26.4, 95% CI 2-sided [-54.1 to 5.8] — Treatment group minus placebo
Statistical Analysis 12: Comparison: A&D - S3 vs Placebo - S3; B/Brisbane; Test type: Superiority; Treatment Difference in Seroconversion R = -8.4, 95% CI 2-sided [-45.4 to 30.5] — Treatment group minus placebo

4. Secondary Outcome: Percentage of Participants With Seroconversion at Day 56 After Vaccination, by Vitamin A Levels at Screening
Description: Secondary analyses will examine sero-conversion based on antibody functions (HAI or neutralization) defined as antibody titers of <1:40 converting to ≥1:40, or a four-fold increase in titer for participants with a starting titer of ≥1:40. Sero-conversion rate (expressed as percentage) will be estimated with 95% confidence interval for participants sufficient and insufficient in vitamin A at screening.
Time Frame: Day 56 after vaccination
Population: Subjects with complete HAI data at day 56. Subjects without a day 56 sample were not included in analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- A&D-S1 VAS: Sub-group of subjects from the A&D-S1 group, vitamin A sufficient (VAS), who received influenza virus vaccine plus vitamin A and D supplements in 2015-16 season
- Placebo-S1 VAS: Sub-group of subjects from the Placebo-S1 group, vitamin A sufficient (VAS), who received influenza virus vaccine plus matched placebo in 2015-16 season
- A&D-S2 VAS: Sub-group of subjects from the A&D-S2 group, vitamin A sufficient (VAS), who received influenza virus vaccine plus vitamin A and D supplements in 2016-17 season
- Placebo-S2 VAS: Sub-group of subjects from the Placebo-S2 group, vitamin A sufficient (VAS), who received influenza virus vaccine plus matched placebo in 2016-17 season
- A&D-S3 VAS: Sub-group of subjects from the A&D-S3 group, vitamin A sufficient (VAS), who received influenza virus vaccine plus vitamin A and D supplements in 2017-18 season
- Placebo-S3 VAS: Sub-group of subjects from the Placebo-S3 group, vitamin A sufficient (VAS), who received influenza virus vaccine plus matched placebo in 2017-18 season
- A&D-S1 Non-VAS: Sub-group of subjects from the A&D-S1 group, vitamin A insufficient/deficient (non-VAS), who received influenza virus vaccine plus vitamin A and D supplements in 2015-16 season
- Placebo-S1 Non-VAS: Sub-group of subjects from the Placebo-S1 group, vitamin A insufficient/deficient (non-VAS), who received influenza virus vaccine plus matched placebo in 2015-16 season
- A&D-S2 Non-VAS: Sub-group of subjects from the A&D-S2 group, vitamin A insufficient/deficient (non-VAS), who received influenza virus vaccine plus vitamin A and D supplements in 2016-17 season
- Placebo-S2 Non-VAS: Sub-group of subjects from the Placebo-S2 group, vitamin A insufficient/deficient (non-VAS), who received influenza virus vaccine plus matched placebo in 2016-17 season
- A&D-S3 Non-VAS: Sub-group of subjects from the A&D-S3 group, vitamin A insufficient/deficient (non-VAS), who received influenza virus vaccine plus vitamin A and D supplements in 2017-18 season
- Placebo-S3 Non-VAS: Sub-group of subjects from the Placebo-S3 group, vitamin A insufficient/deficient (non-VAS), who received influenza virus vaccine plus matched placebo in 2017-18 season
Arm/Group | A&D-S1 VAS | Placebo-S1 VAS | A&D-S2 VAS | Placebo-S2 VAS | A&D-S3 VAS | Placebo-S3 VAS | A&D-S1 Non-VAS | Placebo-S1 Non-VAS | A&D-S2 Non-VAS | Placebo-S2 Non-VAS | A&D-S3 Non-VAS | Placebo-S3 Non-VAS
Number analyzed (Participants) | 2 | 2 | 11 | 11 | 7 | 8 | 3 | 2 | 10 | 9 | 4 | 6
percentage of participants
  H1N1 | 0 [0 to 0] | 0 [0 to 0] | 81.8 [48.2 to 97.7] | 100 [71.5 to 100] | 100 [59.0 to 100] | 87.5 [47.3 to 99.7] | 0 [0 to 0] | 0 [0 to 0] | 60.0 [26.2 to 87.8] | 88.9 [51.8 to 99.7] | 25.0 [0.6 to 80.6] | 83.3 [35.9 to 99.6]
  H3N2 | 0 [0 to 84.2] | 100 [15.8 to 100] | 72.7 [39.0 to 94.0] | 90.9 [58.7 to 99.8] | 71.4 [29.0 to 96.3] | 37.5 [8.5 to 75.5] | 66.7 [9.4 to 99.2] | 0 [0 to 84.2] | 70.0 [34.8 to 93.3] | 66.7 [29.9 to 92.5] | 75.0 [19.4 to 99.4] | 66.7 [22.3 to 95.7]
  B/Phuket | 0 [0 to 0] | 0 [0 to 0] | 45.5 [16.7 to 76.6] | 72.7 [39.0 to 94.0] | 42.9 [9.9 to 81.6] | 25.0 [3.2 to 65.1] | 0 [0 to 0] | 0 [0 to 0] | 10.0 [0.3 to 44.5] | 33.3 [7.5 to 70.1] | 50.0 [6.8 to 93.2] | 33.3 [4.3 to 77.7]
  B/Brisbane | 0 [0 to 0] | 0 [0 to 0] | 36.4 [10.9 to 69.2] | 63.6 [30.8 to 89.1] | 42.9 [9.9 to 81.6] | 50.0 [15.7 to 84.3] | 0 [0 to 0] | 0 [0 to 0] | 20.0 [2.5 to 55.6] | 44.4 [13.7 to 78.8] | 0.0 [0.0 to 60.2] | 16.7 [0.4 to 64.1]

5. Secondary Outcome: HAI Titers at Day 56 After Vaccination, Overall
Time Frame: Day 56 after vaccination
Population: Subjects with complete HAI data at day 56. Subjects without a day 56 sample were not included in analyses.
Measure: Median (Full Range); unit: titers
Arm/Group | A&D-S1 | Placebo - S1 | A&D - S2 | Placebo - S2 | A&D - S3 | Placebo - S3
Number analyzed (Participants) | 5 | 4 | 21 | 20 | 11 | 14
titers
  H1N1 | 5 [5 to 320] | 5 [5 to 5] | 640 [5 to 2560] | 640 [160 to 2560] | 905 [40 to 5120] | 1280 [80 to 10240]
  H3N2 | 320 [5 to 1280] | 480 [160 to 1280] | 1810 [40 to 20480] | 1093 [5 to 5120] | 640 [80 to 2560] | 960 [5 to 5120]
  B/Phuket | 5 [5 to 80] | 5 [5 to 5] | 5 [5 to 160] | 40 [5 to 320] | 5 [5 to 113.14] | 5 [5 to 160]
  B/Brisbane | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 2560] | 40 [5 to 320] | 5 [5 to 452.55] | 42.5 [5 to 640]

6. Secondary Outcome: HAI Titers at Day 56 After Vaccination, by Vitamin A Levels at Screening
Time Frame: Day 56 after vaccination
Population: Subjects with complete HAI data at day 56. Subjects without a day 56 sample were not included in analyses.
Measure: Median (Full Range); unit: titers
Arm/Group | A&D-S1 VAS | Placebo-S1 VAS | A&D-S2 VAS | Placebo-S2 VAS | A&D-S3 VAS | Placebo-S3 VAS | A&D-S1 Non-VAS | Placebo-S1 Non-VAS | A&D-S2 Non-VAS | Placebo-S2 Non-VAS | A&D-S3 Non-VAS | Placebo-S3 Non-VAS
Number analyzed (Participants) | 2 | 2 | 11 | 11 | 7 | 8 | 3 | 2 | 10 | 9 | 4 | 6
titers
  H1N1 | 5 [5 to 5] | 5 [5 to 5] | 640 [80 to 1280] | 640 [160 to 2560] | 1280 [40 to 5120] | 640 [80 to 10240] | 5 [5 to 320] | 5 [5 to 5] | 640 [5 to 2560] | 640 [160 to 2560] | 640 [640 to 3620.4] | 1920 [1280 to 2560]
  H3N2 | 200 [80 to 320] | 720 [160 to 1280] | 1810 [160 to 20480] | 1280 [160 to 5120] | 2560 [160 to 2560] | 320 [5 to 3620.4] | 320 [5 to 1280] | 480 [320 to 640] | 1545 [40 to 2560] | 640 [5 to 2560] | 400 [80 to 1280] | 1920 [640 to 5120]
  B/Phuket | 42.5 [5 to 80] | 5 [5 to 5] | 5 [5 to 80] | 80 [5 to 320] | 5 [5 to 113.14] | 5 [5 to 160] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 160] | 5 [5 to 80] | 42.5 [5 to 80] | 42.5 [5 to 160]
  B/Brisbane | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 640] | 40 [5 to 320] | 80 [5 to 452.55] | 80 [5 to 640] | 5 [5 to 5] | 5 [5 to 5] | 5 [5 to 2560] | 5 [5 to 320] | 5 [5 to 226.27] | 5 [5 to 320]

ADVERSE EVENTS:
Time Frame: 56 days after the final participant was dosed on Day 0.
Arm/Group | A&D-S1 | Placebo - S1 | A&D - S2 | Placebo - S2 | A&D - S3 | Placebo - S3
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/22 | 0/22 | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/22 | 0/22 | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 5/5 | 2/4 | 6/22 | 6/22 | 4/12 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A&D-S1 (N=5) | Placebo - S1 (N=4) | A&D - S2 (N=22) | Placebo - S2 (N=22) | A&D - S3 (N=12) | Placebo - S3 (N=14)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 3 (4) | 3 (3) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fever (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 1 (1) | 2 (2)
Facial trauma/fractured (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left forearm bruise (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT02649192/Prot_SAP_000.pdf